CLINICAL TRIAL: NCT02239549
Title: A Prospective Randomized Study Comparing Jumbo Cold Biopsy Forceps Versus Cold Snare for the Resection of Small Colonic Polyps
Brief Title: Biopsy Forceps Versus Cold Snare for the Resection of Small Colonic Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego Veterans Healthcare System (U.S. Federal Agency)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dr. Mary Krinsky, Clinical Professor of Medicine, San Diego Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H130473; 090012 (Other: UCSD Human Research Protections Program)
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Colonic Polyps
Keywords: Colonic Polyps; Polypectomy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jumbo cold forceps polypectomy group (Experimental): Polypectomy conducted with jumbo cold forceps
  Interventions: Device: Jumbo cold forceps polypectomy
- Cold snare polypectomy group (Experimental): Polypectomy conducted with cold snare
  Interventions: Device: Cold snare polypectomy

INTERVENTIONS:
Device: Jumbo cold forceps polypectomy — The specific jumbo cold forceps used are the Olympus EndoJaw Biopsy Forceps (open jaw diameter 8.5 mm) and the Boston Scientific RJ4 Biopsy Forceps (open jaw diameter 8.8 mm).
  Arms: Jumbo cold forceps polypectomy group
Device: Cold snare polypectomy — The specific cold snares used are the Boston Scientific Captiflex Extra Small Oval Flexible Snare (loop width 11 mm), the US Endoscopy Dsnare Dimunitive Polypectomy and Suction System (loop width 9 mm), or the Boston Scientific Sensation Short Throw Oval Flexible Snare (loop width of 13 mm, 27 mm, or 30 mm).
  Arms: Cold snare polypectomy group

SUMMARY:
The purpose of this study is to evaluate and compare the incomplete resection rates for small colon polyps less than or equal to 6 mm in size using two conventional polypectomy tools, jumbo cold biopsy forceps and cold snare.

DETAILED DESCRIPTION:
The study is a prospective, randomized controlled study involving outpatients undergoing routine colonoscopy. The study is conducted at two academic medical centers, the Veterans Affairs (VA) San Diego Healthcare System and the University of California San Diego (UCSD) Thornton Hospital. Written informed consent is obtained from all participants prior to any study related procedures. Upon enrollment, each patient is randomized via a computer generated randomization scheme to a polypectomy device, either jumbo cold biopsy forceps or cold snare. The randomly allocated polypectomy device is used for polyp resection for polyps less than or equal to 6 mm in size.

All patients undergo standard bowel preparation with 4 liters of polyethylene glycol solution for routine colonoscopy. All colonoscopies are performed using standard colonoscopes (Olympus CF/PCF 160, CF/PCF 180, H-CF/H-PCF 180). Polypectomy tools used are: Olympus Biopsy Forceps, Boston Scientific RJ4 Biopsy Forceps, Boston Scientific Captiflex Extra Small Oval Flexible Snare, US Endoscopy Dsnare Dimunitive Polypectomy and Suction System, and the Boston Scientific Sensation Short Throw Oval Flexible Snare. For all polyps less than or equal to 6 mm in size, documentation of polyp size and anatomic location is conducted.

The jumbo capacity cold forceps polypectomy technique is performed via the following method: After inspection of the polyp, one or more biopsies are taken of the polyp followed by retrieval of the specimens directly from the biopsy forceps. Thereafter, the polypectomy site is vigorously irrigated and visually inspected for evidence of residual polypoid tissue. If residual polypoid tissue is suspected, additional biopsies are taken until the site is considered devoid of polypoid tissue. The total number of bites required for visual completion of polypectomy is recorded.

The cold snare polypectomy technique is performed via the following method: After inspection of the polyp, the snare is used to encircle the polyp with a few millimeter rim of surrounding normal mucosa. The cold snare is used to mechanically transect the polyp without tenting. Thereafter, the resected polyp specimen is suctioned through the colonoscope channel into a trap and retrieval is documented. Next, the polypectomy site is vigorously irrigated and visually inspected for evidence of residual polypoid tissue. If polypoid tissue is still suspected, additional snare excision is performed. The total number of snare excisions required for visual completion of polypectomy is recorded.

For both polypectomy methods, after polyp removal is considered complete, the base and perimeter of the polypectomy site is sampled with a jumbo capacity biopsy forceps with one to three additional biopsies to evaluate for the presence of residual polypoid tissue. All pathology results for the polyp specimens and the polypectomy base specimens are interpreted by a group of VA or UCSD affiliated pathologists.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 80 years
* Undergoing routine colonoscopy

Exclusion Criteria:

* Inflammatory bowel disease
* Cognitive impairment
* Pregnancy
* Presence of a coagulation disorder
* Use of anticoagulant, antiplatelet, or non-steroidal anti-inflammatory drug therapy during the 1 week prior to colonoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2009-04; Primary Completion 2012-05 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Incomplete resection rate | One week after colonoscopy date (when pathology results are available)
  Resected polyp tissue is collected in a unique specimen jar. Tissue from the perimeter and base of the polyp resection site is collected in separate specimen jar. Histological examination by the pathologist is conducted.
  Incomplete resection rate = Number of polyps with residual polyp tissue present in biopsy of the perimeter and base of the polypectomy resection site / Total number of polyps This is calculated for polypectomies utilizing either jumbo capacity biopsy forceps or cold snare.

SECONDARY OUTCOMES:
Rate of tissue retrieval | 1 day (At time of colonoscopy)
  Documentation of whether resected polyp tissue is actually retrieved for placement into specimen jar.
  Rate of tissue retrieval = Number of effectively retrieved polyps for placement into specimen jar / Total number of resected polyps
Rate of procedure-related complications | 1 day (At time of colonoscopy)
  The two procedure related complications that were specifically assessed were post-polypectomy bleeding or perforation.
  Rate of procedure-related complications = Number of colonoscopies with complication of post-polypectomy bleeding or perforation / Total number of colonoscopies

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lee Krinsky, D.O., Principal Investigator — San Diego Veterans Affairs Health Care System
Locations (1):
- Veterans Affairs San Diego Healthcare System, San Diego, California, United States

REFERENCES:
- [Background] Pohl H, Srivastava A, Bensen SP, Anderson P, Rothstein RI, Gordon SR, Levy LC, Toor A, Mackenzie TA, Rosch T, Robertson DJ. Incomplete polyp resection during colonoscopy-results of the complete adenoma resection (CARE) study. Gastroenterology. 2013 Jan;144(1):74-80.e1. doi: 10.1053/j.gastro.2012.09.043. Epub 2012 Sep 25. PMID 23022496
- [Background] Church JM. Clinical significance of small colorectal polyps. Dis Colon Rectum. 2004 Apr;47(4):481-5. doi: 10.1007/s10350-003-0078-6. Epub 2004 Mar 4. PMID 14994108
- [Background] Kapsoritakis AN, Potamianos SP, Koukourakis MI, Tzardi M, Mouzas IA, Roussomoustakaki M, Alexandrakis G, Kouroumalis EA. Diminutive polyps of large bowel should be an early target for endoscopic treatment. Dig Liver Dis. 2002 Feb;34(2):137-40. doi: 10.1016/s1590-8658(02)80244-4. PMID 11926558
- [Background] Efthymiou M, Taylor AC, Desmond PV, Allen PB, Chen RY. Biopsy forceps is inadequate for the resection of diminutive polyps. Endoscopy. 2011 Apr;43(4):312-6. doi: 10.1055/s-0030-1256086. Epub 2011 Mar 16. PMID 21412704
- [Background] Jung YS, Park JH, Kim HJ, Cho YK, Sohn CI, Jeon WK, Kim BI, Sohn JH, Park DI. Complete biopsy resection of diminutive polyps. Endoscopy. 2013 Dec;45(12):1024-9. doi: 10.1055/s-0033-1344394. Epub 2013 Aug 6. PMID 23921846
- [Background] Lee CK, Shim JJ, Jang JY. Cold snare polypectomy vs. Cold forceps polypectomy using double-biopsy technique for removal of diminutive colorectal polyps: a prospective randomized study. Am J Gastroenterol. 2013 Oct;108(10):1593-600. doi: 10.1038/ajg.2013.302. Epub 2013 Sep 17. PMID 24042189
- [Background] Liu S, Ho SB, Krinsky ML. Quality of polyp resection during colonoscopy: are we achieving polyp clearance? Dig Dis Sci. 2012 Jul;57(7):1786-91. doi: 10.1007/s10620-012-2115-6. Epub 2012 Mar 30. PMID 22461018
- [Background] Woods A, Sanowski RA, Wadas DD, Manne RK, Friess SW. Eradication of diminutive polyps: a prospective evaluation of bipolar coagulation versus conventional biopsy removal. Gastrointest Endosc. 1989 Nov-Dec;35(6):536-40. doi: 10.1016/s0016-5107(89)72906-0. PMID 2689263
- [Background] Elmunzer BJ, Higgins PD, Kwon YM, Golembeski C, Greenson JK, Korsnes SJ, Elta GH. Jumbo forceps are superior to standard large-capacity forceps in obtaining diagnostically adequate inflammatory bowel disease surveillance biopsy specimens. Gastrointest Endosc. 2008 Aug;68(2):273-8; quiz 334, 336. doi: 10.1016/j.gie.2007.11.023. Epub 2007 Dec 26. PMID 18155204
- [Background] Draganov PV, Chang MN, Alkhasawneh A, Dixon LR, Lieb J, Moshiree B, Polyak S, Sultan S, Collins D, Suman A, Valentine JF, Wagh MS, Habashi SL, Forsmark CE. Randomized, controlled trial of standard, large-capacity versus jumbo biopsy forceps for polypectomy of small, sessile, colorectal polyps. Gastrointest Endosc. 2012 Jan;75(1):118-26. doi: 10.1016/j.gie.2011.08.019. PMID 22196811
- [Background] Deenadayalu VP, Rex DK. Colon polyp retrieval after cold snaring. Gastrointest Endosc. 2005 Aug;62(2):253-6. doi: 10.1016/s0016-5107(05)00376-7. PMID 16046990
- [Background] Ichise Y, Horiuchi A, Nakayama Y, Tanaka N. Prospective randomized comparison of cold snare polypectomy and conventional polypectomy for small colorectal polyps. Digestion. 2011;84(1):78-81. doi: 10.1159/000323959. Epub 2011 Apr 14. PMID 21494037
- [Background] Komeda Y, Suzuki N, Sarah M, Thomas-Gibson S, Vance M, Fraser C, Patel K, Saunders BP. Factors associated with failed polyp retrieval at screening colonoscopy. Gastrointest Endosc. 2013 Mar;77(3):395-400. doi: 10.1016/j.gie.2012.10.007. Epub 2012 Dec 1. PMID 23211749
- [Background] Tappero G, Gaia E, De Giuli P, Martini S, Gubetta L, Emanuelli G. Cold snare excision of small colorectal polyps. Gastrointest Endosc. 1992 May-Jun;38(3):310-3. doi: 10.1016/s0016-5107(92)70422-2. PMID 1607081
- [Background] Repici A, Hassan C, Vitetta E, Ferrara E, Manes G, Gullotti G, Princiotta A, Dulbecco P, Gaffuri N, Bettoni E, Pagano N, Rando G, Strangio G, Carlino A, Romeo F, de Paula Pessoa Ferreira D, Zullo A, Ridola L, Malesci A. Safety of cold polypectomy for <10mm polyps at colonoscopy: a prospective multicenter study. Endoscopy. 2012 Jan;44(1):27-31. doi: 10.1055/s-0031-1291387. Epub 2011 Nov 28. PMID 22125197